CLINICAL TRIAL: NCT04038723
Title: Proteomic Evaluation of High-Intensity Interval Training Effects on Cardiac Fibrosis
Brief Title: Effects of Interval Training Effects on Cardiac Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 103-7333A3
Record Dates: First submitted 2019-06-18; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-06

CONDITIONS: Fibrosis Myocardial
Keywords: Fibrosis; Ventricle Remodeling; Exercise Training; Proteomics
MeSH Terms: conditions — Fibrosis; Ventricular Remodeling | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre- and Post-HIIT (Experimental): Participants will be evaluated before and after exercise training.
  Interventions: Behavioral: High-intensity interval training

INTERVENTIONS:
Behavioral: High-intensity interval training — Cardiac patients have completed 36 times of exercise training with the exercise frequency of 2-3 times per week. Subjects performed five 3-minute intervals at 80% of VO2peak and each interval was separated by 3-minute exercise at 40% of VO2peak after the warm-up period. The exercise session was terminated by 3-minute cool-down at 30% of VO2peak.

SUMMARY:
The study aimed to highlight the effect of high-intensity interval training (HIIT) on cardiac fibrosis in cardiac patients. From 2009-2018, cardiac patients with measurements of VO2peak, b-type natriuretic peptide, quality of life questionnaire, cardiovascular magnetic resonance imaging with late gadolinium enhancement (CMR-LGE), and preserved serum before and after 36 times of HIIT were enrolled. The human cardiac fibroblast (CF) isolated from human adult ventricle is treated with sera before and after HIIT. Measurements of cell migration as well as cell proliferation and global cell protein profiles before and after HIIT will be performed.

DETAILED DESCRIPTION:
From January 1, 2009 to December 31, 2018, cardiac patients with stable clinical status for greater than 4 weeks have completed 36 times of HIIT. Subjects with clinical assessments (listed below) before and after HIIT will be included.

*Baseline information, including age, gender, body mass index, duration disease duration, co-morbidities and medication history were reviewed. Subjects with echocardiographic examination, short form-36 health survey (SF-36) for qualities of life, graded cardiopulmonary exercise test (CPET), cardiac magnetic resonance imaging with late gadolinium enhancement (CMR-LGE), blood chemistry tests (hematocrit, brain natriuretic peptide, high-sensitivity C-reactive protein, creatinine), and preserved sera before and after HIIT.*

Cell behaviors Human cardiac fibroblast (CF) isolated from human adult ventricle (HCF-av cell, ScienCell Research Laboratories, Carlsbad, CA, USA) are cultured in medium containing 10 % FBS, 1% fibroblast growth supplement, and 1% penicillin/streptomycin. Cells (1x10^5) were seeded in dishes of 10-cm diameter and were cultured in the above medium overnight. We used 10% of the patient serum in substitution for the 10% fetal bovine serum (FBS) to treat human cardiac fibroblast (CF) isolated from human adult ventricle (HCF-av cell, ScienCell Research Laboratories, Carlsbad, CA, USA), and serum effects on CF were evaluated.

Cell Culture Human cardiac fibroblasts (CFs) isolated from human adult ventricle (HCF-av cell, ScienCell Research Laboratories, Carlsbad, CA, USA) were cultured in medium containing 10 % FBS, 1% fibroblast growth supplement, and 1% penicillin/streptomycin. Cells (1x10^5) were seeded in dishes of 10-cm diameter and were cultured in the above medium overnight.

Cell migration assay The cell migration speed in the serum obtained from cardiac patients pre- and post-HIIT was determined as described previously. In brief, HCF-av cells of 3000 were plated on each 3.5-cm Petri dishes with polyacrylamide substrates and were harvest in media containing 10% of cardiac patient sera before and after HIIT. Phase contrast images were recorded using a cooled charge-coupled device camera (Photometrics, Tucson, AZ), attached to an Eclipse Ti-E inverted microscope system (Nikon Instruments Inc., Melville, NY) equipped with a 20X, numerical aperture 0.75 Achromat phase objective lens and a INU series stage top incubator (Tokai HIT Co., Ltd., Shizuoka-ken, Japan). The position of the cell was determined every 10 min for a period of 120-180 mins, based on the center of the nucleus. Migration speed was calculated based on the persistent random walk equation.

Cell proliferation assay HCF-av cells of 7.5x10^3 were plated in each well (0.95 cm^2 growth area) of a 48-well cell culture plate (Sigma-Aldrich, St. Louis, MO) with ordinary medium for 8 hours. They were then cultured in a starvation medium containing 1.5% FBS overnight. The prepared cells were stained with Hoechst 33342 (Thermo Fisher Scientific Inc., Waltham, MA) for 15 mins and were then washed twice in phosphate buffered saline. They were separately treated with 10% FBS (10 wells), and 10% patient serum obtained from our subjects before (24 wells) and after HIIT (24 wells). We used IN Cell Analyzer 1000 cellular imaging and analysis system (GE Healthcare Bio-Science Corp., Piscataway, NJ) to count cell numbers at 0, 24 hours, and 48 hours after harvested with the three different culture media.

Proteomic analysis Protein concentrations of different treatment groups were determined by Bicinchoninic acid assay (ThermoFisher Scientific Inc.). Protein mixtures were separated by electrophoresis on 12.5% SDS-PAGE gel followed by in-gel enzyme digestion according to the following procedure. After thermal denaturation at 95 oC for 5 min, protein samples were reduced through the addition of dithiothreitol (DTT) to a ﬁnal concentration of 10 mM and incubated at 50 oC for 30 min. Alkylation was performed by adding iodoacetamide (IAA) to a ﬁnal concentration of 20 mM prior to incubation at room temperature for 30 min in the dark. A second aliquot of DTT was then added to quench unreacted IAA. For trypsin digestion, trypsin was added (1:50, w/w) and the reaction mixture was incubated at 37 oC for 12 h. The trypsin digestion was quenched through the addition of a 10 microL formic acid (10%). Digested peptides were dried by speedvac for mass analysis.

The tryptic peptides were analyzed on a LTQ-FT (linear quadrupole ion trap-Fourier transform ion cyclotron resonance) hybrid mass spectrometer (Thermo Fisher Scientific, Inc., Waltham, MA) equipped with a nano-electrospray ion source (New Objective, Inc., Woburn, MA) in positive ion mode. The liquid chromatography system was the Agilent 1100 Series HPLC (Agilent Technologies, Palo Alto, CA) with the Famos autosampler (LC Packings, San Francisco, CA). Peptide solution was injected onto a self-packed precolumn (150 microm I.D. x 20 mm, 5 microm, 200 Å) and the chromatographic separation was sequentially performed on a self-packed reversed phase C18 nano-column (75 microm I.D. x 300 mm, 5 microm, 100 Å) by using 0.1% formic acid in water (mobile phase A) and 0.1% formic acid in 80% acetonitrile (mobile phase B). A linear gradient from 5 to 40% mobile phase B for 40 min at a flow rate of 300 nL/min was applied. Electrospray voltage was applied at 2.0 kV and capillary temperature was set at 200 oC. A scan cycle was initiated with a full-scan survey MS spectrum (m/z 300 - 2000) performed on the FT-ICR mass spectrometer with resolution of 100,000 at 400 Da. Ten most abundant ions detected in this scan were subjected to a MS/MS experiment performed in the linear quadrupole ion trap (LTQ) mass spectrometer. Ion accumulation (Auto Gain Control target number) and maximal ion accumulation time for full-scan and MS/MS were set at 1 x 106 ions, 1000 ms and 5 x 104 ions, 200 ms. Ions were fragmented by use of CID (collision induced dissociation) with the normalized collision energy was set to 35 %, activation Q was 0.3 and activation time was 30 ms.

All experiment RAW files were subjected to MaxQuant (1.5.3.30) for the label-free protein quantitation. The variable post-translational modifications of search parameters in MaxQuant were assigned to include the oxidation of methionine, and the phosphorylation of serine/threonine/tyrosine. The carbamidomethylation of cysteine was assigned as the fixed modification. The enzyme for digestion was assigned to be trypsin with the miss cleavage number two. Homo Sapiens protein sequences from SwissProt 2018_06 were used for MS/MS search. Protein quantitation results were obtained by the LFQ intensity from MaxQuant.

Statistical analysis Wilcoxon matched-pairs signed-ranks test was used to compare exercise capacity parameters, CMR-LGE results, blood chemistry data, and SF-36 scores before and after HIIT in each individual. Student t test was used to assess protein level changes before and after HIIT.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients, diagnosed according to the Framingham heart failure diagnostic criteria, with stable clinical status for greater than 4 weeks after conservative treatment or intervention were enrolled in the study.

Exclusion Criteria:

Those who were

* < 20 years
* under anti-coagulant therapy
* unable to exercise > 1 year owing to non-cardiovascular disease
* pregnant or plan to be pregnant within one year
* plan to have cardiac transplant within 6 months
* uncorrected valvular heart disease related heart failure
* congenital heart disease related heart failure
* Other exercise contraindications：

  1. unstable angina
  2. resting systolic blood pressure> 200 mmHg or resting diastolic blood pressure> 110 mmHg
  3. orthostatic blood pressure drop (systolic blood pressure drop > 20 mmHg)。
  4. critical aortic stenosis stenosis (peak systolic pressure gradient> 50 mmHg and aortic valve opening < 0.75 cm2)。
  5. acute fever
  6. uncontrolled uncontrolled atrial or ventricular dysrhythmias
  7. uncompensated congestive heart failure
  8. 3-degree AV block)
  9. acute pericarditis and/or myocarditis
  10. recent embolism < 6 months
  11. thrombophlebitis
  12. restin ST segment displacement > 2mm
  13. patients with uncontrolled diabetes (resting serum glucose > 300mg/dL or > 250mg/dL with ketone body) was excluded in the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Cardiac output (CO) | 3-4 months (for 36 times of exercise training)
  Cardiac output in milliliter per minute measured by cardiac magnetic resonance imaging with late gadolinium enhancement before and after exercise training
Cardiac mass | 3-4 months (for 36 times of exercise training)
  Cardiac mass in gram measured by cardiac magnetic resonance imaging with late gadolinium enhancement before and after exercise training
Left ventricular end-systolic volume (LVESV) | 3-4 months (for 36 times of exercise training)
  LVESV in milliliter measured by cardiac magnetic resonance imaging with late gadolinium enhancement before and after exercise training
Left ventricular end-diastolic volume (LVEDV) | 3-4 months (for 36 times of exercise training)
  LVEDV in milliliter measured by cardiac magnetic resonance imaging with late gadolinium enhancement before and after exercise training
Extracellular volume fraction (ECV) | 3-4 months (for 36 times of exercise training)
  ECV in percent (%) measured by cardiac magnetic resonance imaging with late gadolinium enhancement before and after exercise training
Proteomics | 3-4 months (for 36 times of exercise training)
  Protein level changes in fold change in cardiac fibroblast before and after exercise training

SECONDARY OUTCOMES:
Peak exercise capacity (VO2peak) | 3-4 months (for 36 times of exercise training)
  VO2peak in ml/min/kg measured by cardiopulmonary function test before and after exercise training
Peak cardiac output (CO) | 3-4 months (for 36 times of exercise training)
  Peak CO in millimeter per minute measured by non-invasive cardiac output measurement during exercise test before and after exercise test
Oxygen uptake efficiency slope (OUES) | 3-4 months (for 36 times of exercise training)
  OUES in liter per minute/log(Liter per minute) derived from oxygen consumptions along time during exercise test before and after exercise test
Ventilation/VCO2 ratio (Ve-VCO2) | 3-4 months (for 36 times of exercise training)
  Ve-VCO2, a number, derived from exhaled CO2 (ml/min/kg) versus ventilation (ml/min/kg) graph along time during exercise test before and after exercise test
Migration speed | 3-4 months (for 36 times of exercise training)
  Cell migration speed in micrometer per minute of cardiac fibroblast measured before and after exercise training
Cell proliferation curve | 3-4 months (for 36 times of exercise training)
  Cell proliferation curve of cardiac fibroblasts in numbers (at initial state, 24 hours after incubation, and 48 hours after incubation) measured before and after exercise training
Hematocrit (Hct) | 3-4 months (for 36 times of exercise training)
  Hct in percent (%) from blood chemistry study before and after exercise training
Brain natriuretic peptide (BNP) | 3-4 months (for 36 times of exercise training)
  BNP in picogram per milliliter from blood chemistry study before and after exercise training
High-sensitivity C-reactive protein (hsCRP) | 3-4 months (for 36 times of exercise training)
  hsCRP in milligram per liter from blood chemistry study before and after exercise training
Creatinine (Cre) | 3-4 months (for 36 times of exercise training)
  Cre in milligram per deciliter from blood chemistry study before and after exercise training
Physical component score (PCS) | 3-4 months (for 36 times of exercise training)
  Physical role function obtained from short form 36 questionnaire (SF-36) before and after exercise training. The SF-36 consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Mental component score (MCS) | 3-4 months (for 36 times of exercise training)
  Mental health score obtained from short form 36 questionnaire (SF-36) before and after exercise training. The SF-36 consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu CC, Wang JS, Shyu YC, Fu TC, Juan YH, Yuan SS, Wang CH, Yeh CH, Liao PC, Wu HY, Hsu PH. Hypermethylation of ACADVL is involved in the high-intensity interval training-associated reduction of cardiac fibrosis in heart failure patients. J Transl Med. 2023 Mar 10;21(1):187. doi: 10.1186/s12967-023-04032-7. PMID 36894992